# **DISCLOSURE**

#### REDACTED STATISTICAL ANALYSIS PLAN AMENDMENT

#### MEDI4736-NHL-001

# A PHASE 1/2, OPEN LABEL, MULTICENTER STUDY TO ASSESS THE SAFETY AND TOLERABILITY OF DURVALUMAB (ANTI-PD-L1 ANTIBODY) AS MONOTHERAPY AND IN COMBINATION THERAPY IN SUBJECTS WITH LYMPHOMA OR CHRONIC LYMPHOCYTIC LEUKEMIA

The "FUSION NHL-001" Study

The information contained in the attached report is the property of Celgene and should **not be** shared or used for any purpose other than that for which it was provided.

Celgene is committed to providing information about its clinical trials to researchers and patients with the goal of furthering science and enhancing healthcare worldwide. Laws and regulations require, however, that Celgene protects patient privacy. The company may further have legal or contractual obligations not to disclose commercial or technical information provided by or related to certain partner companies or vendors.

The attached report is presented in its original format, but certain information has been redacted in order to comply with the aforementioned obligations or to protect Celgene's confidential commercial information. The redactions are based on the following principles:

- Redacted information has been replaced by grey space, maintaining original spacing and pagination.
- Any information that might allow the identification of individuals has been redacted for anonymization.
- Attachments to this report that contain confidential information are not made available. Such
  attachments include those that contain identifiable patient information, such as subject listings,
  narratives, and profiles. They also may contain confidential commercial information such as
  methodologies, and hypothesis generating and exploratory analyses.
- Cross-references to these attachments (such as links to subject listings in Section 16.2) are not redacted from the body of the report. However, the hyperlinks in the electronic document are no longer functional.
- Information about Celgene vendors and their services are redacted because many contracts prohibit disclosure of that information. Further, laws and regulations prevent us from disclosing certain information about our vendors or their services because it is protected by copyright.

Information about Celgene's redaction policies and the availability of additional data from this report may be found at http://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/.

# STATISTICAL ANALYSIS PLAN AMENDMENT 1

A PHASE 1/2, OPEN-LABEL, MULTICENTER STUDY TO ASSESS THE SAFETY AND TOLERABILITY OF DURVALUMAB (ANTI-PD-L1 ANTIBODY) AS MONOTHERAPY AND IN COMBINATION THERAPY IN SUBJECTS WITH LYMPHOMA OR CHRONIC LYMPHOCYTIC LEUKEMIA

STUDY DRUG: MEDI4736

PROTOCOL NUMBER: MEDI4736-NHL-001

FINAL PROTOCOL DATE: 06 Nov 2015

PROTOCOL AMENDMENT No. 1 04 May 2017

DATE:

PROTOCOL AMENDMENT No 2 14 Dec 2017

**DATE:** 

Prepared by:
ICON Clinical Research
On behalf of
Celgene International II Sarl
Rue des Moulins 4
2108 Couvet
Switzerland

#### CONFIDENTIAL

The information contained in this document is regarded as confidential and, except to the extent necessary to obtain informed consent, may not be disclosed to another party unless such disclosure is required by law or regulations. Persons to whom the information is disclosed must be informed that the information is confidential and may not be further disclosed by them

# SIGNATURE PAGE

| SAP TITLE MEDI4736-NHL-001 Statistical Analysis Plan SAP VERSION, DATE Version 2.0 (Amendment 1), 23 Apr 2019 SAP AUTHOR A Phase 1/2, open-label, multicenter study to assess the safety and tolerability of durvalumab (anti-PD-L1 antibody) as monotherapy and in combination therapy in subjects with lymphoma or chronic lymphocytic leukemia INVESTIGATIONAL PRODUCT PROTOCOL NUMBER MEDI4736-NHL-001 PROTOCOL VERSION, DATE SIGNATURE SIGNATURE SIGNATURE STATEMENT By my signature, 1 indicate 1 have reviewed this SAP and find its contents to be acceptable. Statistical Therapeutic Area Hand Signature |
|---|
| SAP VERSION, DATE Version 2.0 (Amendment 1), 23 Apr 2019 A Phase 1/2, open-label, multicenter study to assess the safety and tolerability of durvalumab (anti-PD-L1 antibody) as monotherapy and in combination therapy in subjects with lymphoma or chronic lymphocytic leukemia INVESTIGATIONAL PRODUCT PROTOCOL NUMBER MEDI4736 PROTOCOL VERSION, DATE SIGNATURE SIGNATURE SIGNATURE By my signature, 1 indicate I have reviewed this SAP and find its contents to be acceptable. Statistical Therapeutic Area Hand |
| PROTOCOL TITLE A Phase 1/2, open-label, multicenter study to assess the safety and tolerability of durvalumab (anti-PD-L1 antibody) as monotherapy and in combination therapy in subjects with lymphoma or chronic lymphocytic leukemia INVESTIGATIONAL PRODUCT PROTOCOL NUMBER MEDI4736 PROTOCOL VERSION, DATE By my signature, 1 indicate 1 have reviewed this SAP and find its contents to be acceptable. Statistical Therapeutic Area Hand |
| A Phase 1/2, open-label, multicenter study to assess the safety and tolerability of durvalumab (anti-PD-L1 antibody) as monotherapy and in combination therapy in subjects with lymphoma or chronic lymphocytic leukemia INVESTIGATIONAL MEDI4736 PROTOCOL NUMBER MEDI4736-NHL-001 PROTOCOL VERSION, Amendment No. 2, 14 Dec 2017 DATE SIGNATURE By my signature, 1 indicate I have reviewed this SAP and find its contents to be acceptable. Statistical Therapeutic Area Hand |
| PROTOCOL TITLE durvalumab (anti-PD-L1 antibody) as monotherapy and in combination therapy in subjects with lymphoma or chronic lymphocytic leukemia INVESTIGATIONAL PRODUCT PROTOCOL NUMBER MEDI4736 PROTOCOL VERSION, DATE SIGNATURE By my signature, 1 indicate 1 have reviewed this SAP and find its contents to be acceptable. Statistical Therapeutic Area Head |
| PRODUCT PROTOCOL NUMBER MEDI4736-NHL-001 PROTOCOL VERSION, DATE SIGNATURE By my signature, 1 indicate 1 have reviewed this SAP and find its contents to be statistical Therapeutic Area Hand |
| PROTOCOL VERSION, DATE SIGNATURE By my signature, 1 indicate I have reviewed this SAP and find its contents to be STATEMENT Statistical Therapeutic Area Hand |
| SIGNATURE SIGNATURE By my signature, I indicate I have reviewed this SAP and find its contents to be STATEMENT acceptable. Statistical Therapeutic Area Head |
| STATEMENT acceptable. Statistical Therapeutic Area Hand |
| Signature |
| Printed Name |
| Lead Clinical Resear |
| Signature |
| Printed Name |
| Lead Product Safety Physician |
| Signature |
| Printed Name Date |

# **SIGNATURE PAGE**

| | SIGNATURE PAGE |
|---|---|
| STATISTICAL ANALYSIS PLAN (SAP) AND SAP AMENDMENT APPROVAL SIGNATURE PAGE | |
| SAP TITLE | MEDI4736-NHL-001 Statistical Analysis Plan |
| SAP VERSION, DATE | Version 2.0 (Amendment 1), 23 Apr 2019 |
| SAP AUTHOR | |
| PROTOCOL TITLE | A Phase 1/2, open-label, multicenter study to assess the safety and tolerability of durvalumab (anti-PD-L1 antibody) as monotherapy and in combination therapy in subjects with lymphoma or chronic lymphocytic leukemia |
| INVESTIGATIONAL PRODUCT | MEDI4736 |
| PROTOCOL NUMBER | MEDI4736-NHL-001 |
| PROTOCOL VERSION,<br>DATE | Amendment No. 2, 14 Dec 2017 |
| SIGNATURE<br>STATEMENT | By my signature, I indicate I have reviewed this SAP and find its contents to be acceptable. |
| Statistical Therapeutic Are | a Head |
| Signature | |
| Printed Name | Date |
| Lead Clinical Research | 20. |
| Signature | |
| Printed Name | |
| Lead Product Safety Physi | cian |
| Signature | |
| Printed Name | Date |
| Harry Control of the | |

#### Reason of the amendment

This statistical analysis plan (SAP) amendment details the Efficacy Evaluable Population in the case of subjects do not have a post-baseline response assessment before death.

### **Efficacy Evaluable Population**

Per SAP version 1.0, section 4.2.2, the Efficacy Evaluable Population is defined as follow:

Efficacy Evaluable (EE) Population (for the dose-finding, dose-confirmation, and dose-expansion part) is defined as all subjects who complete at least 1 cycle of their assigned treatment, have baseline, and at least 1 post-baseline tumor response assessment. Subjects will be analyzed according to their initial treatment arm and dose level allocation.

# Changed to

Efficacy Evaluable (EE) Population (for the dose-finding, dose-confirmation, and dose-expansion part) is defined as all subjects who complete at least 1 cycle of their assigned treatment, have baseline, and at least 1 post-baseline tumor response assessment.

A subject who died before Cycle 4 Day 1 (i.e. before the first IWG or IWCLL response assessment scheduled per protocol) and without having done any unscheduled post-baseline IWG or IWCLL response assessment will be included in the Efficacy Evaluable Population.

Subjects will be analyzed according to their initial treatment arm and dose level allocation.

#### Rational:

The first efficacy assessment is performed at Cycle 4 Day 1, any subject who died before and without having done any unscheduled post-baseline IWG or IWCLL response assessment cannot have a post baseline assessment and should not be excluded from the Efficacy Evaluable Population for that criterion.